CLINICAL TRIAL: NCT06775418
Title: Comparison Between Ultrasound Guided Erector Spinae Plane Block and Dexmedotomidine in Lumber Spine Surgeries.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed wagih Ezzat deusouky, lecturer of anasthesia,intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS61/2024
Record Dates: First submitted 2025-01-05; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Analgesia, Postoperative
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group U (Experimental): Group (U) will receive bilateral US guided single shot ESPB, 30 ml of bupivacaine 0.25% on each side after induction of anesthesia.
  Interventions: Procedure: Ultrasound erector spinae plane block
- group D (Experimental): Group (D)will receive the study drug infusion (Dexmedetomidine) after induction of anesthesia.
  Interventions: Procedure: dexamedotomidine infusion after induction of anesthesia

INTERVENTIONS:
Procedure: Ultrasound erector spinae plane block — Patients will be subdivided randomly into two groups (15 patients each) using computer generated random numbers with closed envelopes:
  Group U (15 patients):will receive bilateral US guided single shot ESPB, 30 ml of bupivacaine 0.25% on each side after induction of anesthesia.
  Arms: group U
Procedure: dexamedotomidine infusion after induction of anesthesia — Patients will be subdivided randomly into two groups (15 patients each) using computer generated random numbers with closed envelopes:
  Group D (15 patients):will receive the study drug infusion (Dexmedetomidine) after induction of anesthesia.
  Arms: group D

SUMMARY:
Ultrasound (US) guided Erector spinae plane block (ESPB) as a new trunchal fascial plane block technique was proposed in 2016. US guided ESPB has aroused the interest of many nerve block experts. The goal of this study is to evaluate the effect of US guided ESPB versus (VS) intravenous Dexmedotomidine on postoperative analgesia and intra operative hemodynamic parameters in lumbar spine surgeries.

The aim of this study is to compare the efficacy of ESPB to intravenous Dexmedetomidine in patients who are undergoing elective lumber spine surgeries regarding the effect on postoperative analgesia and intra operative hemodynamic parameters.

DETAILED DESCRIPTION:
The use of US guided ESPB in lumbar spine surgery has not been extensively studied in clinical research. Although there is limited research available, some studies have highlighted differences in the mechanism and effectiveness of the block in different regions of the erector spinae muscle. Some scholars question the practicability of US guided ESPB in lumbar surgery. This suggests that further investigation is needed to understand the practicality and potential benefits of using ultrasound-guided ESPB in lumbar spine surgery.

Dexmedetomidine, a highly selective α₂ receptor agonist, has a sympatholytic, sedative, amnestic and opioid sparing effect. It does not cause respiratory depression and can therefore be used as an adjuvant in certain clinical settings .

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients. aged 18 to 50 years. 70 to 80 kg.

Exclusion Criteria:

* patients under 18 years of age.

  * History of Allergic reactions to study drugs.
  * Opioid or analgesic abuse, and chronic treatment with opioids, or nonsteroidal anti-inflammatory drugs.
  * History of bleeding tendency or coagulopathy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
(VAS) during the 1st 24 hours | 24 HOURS
  Pain will be assessed on admission and at 2, 4, 8, 12 and 24 hours at rest and with passive flexion of hip and knee joint using visual analogue scale (VAS) ranging from 0 for no pain to 10 for worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes